CLINICAL TRIAL: NCT05100576
Title: Randomized Controlled Clinical Trial of Telemedicine-guided Lifestyle Intervention in Diabetic Patients During Intensive Insulin Therapy.
Brief Title: Intensified Insulin Therapy With Telemedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TMED_INZULIN_001
Record Dates: First submitted 2021-10-06; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Intensified Insulin Therapy; Diabetes
Keywords: telemedicine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): This group gets the telemedicine system, with the devices, and gets life-style guide by telephone consultation/ visits, during 3 months
  Interventions: Device: Telemedicine system users
- Comparator group (No Intervention): This group gets the normal, evidence based therapy, without extra visits.

INTERVENTIONS:
Device: Telemedicine system users — Telemonitoring by medical devices connected to a software system with a router.
  Arms: Active group

SUMMARY:
Investigation of the effect of a 3-month telemedicine-led lifestyle intervention in individuals requiring intensified insulin therapy.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the development of HbA1c levels in patients requiring 3 months of intensified insulin therapy using standard therapy and telemedicine devices currently in use.

The telemedicine system contains a mobile phone-based nutrition diary, bluetooth-related wrist activity meter, weight scale, blood pressure monitor, blood glucose meter, and IT system for transmitting and displaying data from these devices.

ELIGIBILITY:
Inclusion Criteria:

* Women or men between the ages of 18 and 75
* Patient with Diabetes who needs intensified insulin therapy HbA1c> = 8%
* IT proficiency is at least basic for cell phones (answering / making a voice call).
* Signing a informed consent
* For women with childbearing potential, by definition, all women who who are physiologically able to conceive are twofold use of contraception
* The subject communicates well with the investigator and is able to perform the test to understand and help comply with the requirements of the protocol

Exclusion Criteria:

* informed refusal any time after the sign of the informed consent
* Planned invasive cardiac intervention (catheter vasodilation or surgical coronary artery bypass grafting, keyboard surgery or replacement)
* Tumor disease
* Pregnant or lactating women
* Any medical condition that does not allow participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c level | 3 months
  Investigation of the effect of a 3-month telemedicine-led lifestyle intervention on HbA1c levels in individuals requiring insulin therapy

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  Safety of the device system
change of hypoglycemic episodes | 3 months
  Number of hypoglycemic episodes
Difference in the decisions between the two type of visits | 3 months
  Consistency of investigators' decisions based on telemedicine data and personal visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No